CLINICAL TRIAL: NCT06954545
Title: Effectiveness of a Role-play Based School Intervention in Primary School Students: a Non-randomized Cluster Controlled Trial
Brief Title: Outcomes of a Game-based Educational Intervention: Healthy Kids
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Lacin Aksoy, Principal investigator, Marmara University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MU-FM-LA-01
Record Dates: First submitted 2025-04-14; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Obesity and Overweight; Child Health; Physical Activity
Keywords: educational intervention; prevention of obesity
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Intervention Model Description: intervention group with healthy kids programme, control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): A training was conducted only once, which did not include play and role play and provided information
- Intervention group (Experimental): Two schools were determined as control and intervention groups. An 8-week interactive-game-based intervention program will be applied to children in the intervention group who are at risk for obesity. The program was shaped by a physician-dietician-psychologist and a professional theater actor physician.
  Interventions: Behavioral: Healthy Kids Programme

INTERVENTIONS:
Behavioral: Healthy Kids Programme — Our intervention was prepared by adopting an interactive curriculum shaped on role-play with visual materials and toy models of foods appropriate for the age of the children
  Arms: Intervention group

SUMMARY:
235 / 5.000 Investigators aimed to reduce the risk of obesity by trying a new intervention method that is role-play based, interactive and fun with age-appropriate play materials, considering that learning through play is more efficient.

DETAILED DESCRIPTION:
It was aimed to reduce the risk of obesity by trying a new intervention method based on role-play, interactive and fun with age-appropriate game materials, considering that learning through play is more efficient.

Two schools were determined as control and intervention groups. An 8-week interactive-game-based intervention program will be applied to children in the intervention group who are at risk for obesity. The program was shaped by a physician-dietician-psychologist and a professional theater actor.

Family Nutrition and Physical Activity (FNPA) score, Food index (FI) score and BMI will be grouped for each child and a risk score will be calculated based on the total score they receive. It will be checked whether there is a decrease in this score after the training.

ELIGIBILITY:
Inclusion Criteria:

* All participants who do not meet the criteria of whether or not they agree to participate in the study will be included in the study.

Exclusion Criteria:

* neurodevelopmental delays
* metabolic disorders potentially leading to obesity
* physical disabilities
* those whose parents or guardians declined participation.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
BMI (body mass index) | All measurements will be collected at 0, 3 and 6 months
  We inputted the height and weight measurements into the WHO( World Health Organization) AntroPlus tool and assessed the BMI z-score. We will group the participants as underweight-normal, overweight, obese and morbidly obese.

SECONDARY OUTCOMES:
FNPA scores | All measurements will be collected at 0, 3 and 6 months
  Researchers will distribute the Family Nutrition and Physical Activity (FNPA) scale to parents. Parents will collect the questionnaires after they complete them. Children who score high on the FNPA scales are thought to have protective family behaviors against obesity. There is no cut-off point for the scale.
FI Scores | All measurements will be collected at 0, 3 and 6 months
  Researchers will collect data by distributing the Food Index to families and collecting it.
  A high score on the Food Index is known to protect against obesity. There is no cut-off point for the index.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu uzuner, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No